CLINICAL TRIAL: NCT01223781
Title: Biofeedback-based Motor Learning to Ameliorate Freezing of Gait
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Meir Plotnik, PhD, Tel Aviv Sourasky Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 510-10-TLV
Record Dates: First submitted 2010-10-17; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Gait; Parkinson Disease
Keywords: Freezing; biofeedback; motor learning; freezing of gait in PD
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Feedforward stimulation (Experimental): Prior to any gait condition likely to invoke freez, auditory stimulation is presented
  Interventions: Behavioral: Biofeedback-based motor learning for PD
- Feedback stimulation (Experimental): Once a device identifies freezing, a auditory stimulation is triggered
  Interventions: Behavioral: Biofeedback-based motor learning for PD

INTERVENTIONS:
Behavioral: Biofeedback-based motor learning for PD — Prior to freezing episodes, auditory stimulation is triggered

SUMMARY:
Objective/Rationale:

The investigators objective is to demonstrate that an intervention program based on motor learning principles can be applied to train subjects with Parkinson's disease (PD) who suffer from freezing to walk in a way that minimizes the occurrence of freezing. Since sufficient motor learning capabilities are preserved in PD, the investigators hypothesize that an intervention program that targets the time periods just prior to an approaching freezing episode can modify the walking strategies so that the episode will now be averted.

Project Description:

The freezing burden will be quantified in subjects with PD before and after 6 weeks of training. Two types of interventions (20 subjects in each group) will be tested: 1) Open-loop group (OLG); 2) Closed-loop group (CLG). Each session of the OLG training includes walking courses aimed at provoking freezing episodes. The experimenter will trigger an auditory rhythmic stimulation (RAS) in walking conditions likely to invoke freezing (e.g., turning) and the subject will learn to synchronize his/her gait with the auditory cues, i.e., to keep the walking pace and coordination and, as a result, to avoid freezing. Similar principles will apply for the CLG training; however, the RAS will be elicited automatically by a device that recognizes an approaching freezing episode.

Relevance to Diagnosis/Treatment of Parkinson's Disease:

If even partially successful, the investigators will show, for the first time that freezing of gait is amenable to motor learning and that appropriate training with external cueing can alleviate these motor blockades. While future studies will be needed to further assess long-term efficacy and other important questions about clinical efficacy and the mechanisms involved, this study should go a long way towards improving the investigators understanding of freezing of gait and its amenability to appropriate therapy.

Anticipated Outcome:

The investigators anticipate that after intensive training, the central nervous system (CNS) of subjects with PD will be able to anticipate impending freezing episodes based on awareness of the environmental conditions (e.g., an approaching turn) and/or based on sub-conscious response to a deteriorating gait pattern. As a result, an automated motor response that paces and coordinates gait will be internally triggered by the CNS and the approaching freezing episode will be averted. The overall freezing burden will therefore decrease in trained subjects.

DETAILED DESCRIPTION:
Overview: This will be a randomized trial to demonstrate the effects of 6-weeks of training with open-loop or triggered, closed-loop cueing. PD+ FOG patients will be studied before and after 6 weeks of training (total of 18 sessions) and one month later (to begin to assess retention). The two intervention groups will receive training sessions designed to enhance implicit motor learning and avoidance of FOG. This will be the first study to assess these novel paradigms. If the results support the hypotheses, further studies will be needed including a placebo-controlled trial. 20 subjects will be included in the feed-forward, open-loop group (OLG) and 20 in the feedback, closed-loop group (CLG) (based on power analysis to provide 80% power at α=0.05). Participants will be recruited on a rolling admission basis (about 2 subjects per week over ~20 weeks) and will be randomly assigned to one of the 2 groups. Pre, post and retention effects will be tested without knowledge of group assignment. A (repeated measures) mixed models statistical approach will be used to evaluate within and across group effects over time, adjusting for baseline values. The study will be conducted under the auspices of the Laboratory for Gait and Neurodynamics and the Movement Disorders Unit (MDU) at the Tel-Aviv Sourasky Medical Center. At all times during training and testing, the subjects will be closely monitored by a research assistant to ensure safety.

ELIGIBILITY:
Inclusion Criteria:1) Have a diagnosis of PD 2) Suffer from the FOG symptom. Subjects must score 2 or more on item #3 of the subjective FOG questionnaire (FOG-Q)and exhibit two or more FOG episodes during a short, functional FOG evaluation procedure that includes FOG-provoking conditions (e.g., turns, doorways) and 5 laps of walking in a figure 8 shaped trajectory 3) Free of serious co-morbidities or acute illness that would make training inappropriate.

Exclusion Criteria:

1) Unable to walk unassisted for at least 5 minutes with ample rest. 2)Brain surgery.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Number of freezing episodes | 3 days
  In lab examinaiton and then in 3 days of ambulatory monitoring, the nubmer of freezing episodes will be counted before and after the intervention.

SECONDARY OUTCOMES:
duration of freezing episodes | 3 days
  In lab examinaiton and then in 3 days of ambulatory monitoring, the duration of freezing episodes will be counted before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for Gait and Neurodynamics, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Bachlin M, Plotnik M, Roggen D, Maidan I, Hausdorff JM, Giladi N, Troster G. Wearable assistant for Parkinson's disease patients with the freezing of gait symptom. IEEE Trans Inf Technol Biomed. 2010 Mar;14(2):436-46. doi: 10.1109/TITB.2009.2036165. Epub 2009 Nov 10. PMID 19906597